CLINICAL TRIAL: NCT01130480
Title: Accu-Chek missiOn: SMBG in Patients With diAbetes on inSulin Study (COMPASS) - Multiple Center, Open, and Non-randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RD000933
Record Dates: First submitted 2010-05-19; First posted 2010-05-26 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (1):
- A (Experimental)
  Interventions: Device: Accu-Chek Integra Glucometer

INTERVENTIONS:
Device: Accu-Chek Integra Glucometer

SUMMARY:
COMPASS is a status and intervention study for the self-monitoring of blood glucose (SMBG) in type 2 diabetic patients with insulin treatment. This multi-centre, open-label prospective study will assess the use and frequency of SMBG and blood glucose control and its influencing factors with the help of Accu-Chek Integra glucometer. Patients with type 2 diabetes mellitus who have received more than 3 months of insulin therapy are eligible to participate in this study. The anticipated duration of the study is 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetes mellitus patients who have received insulin treatment for more than 3 months
* Patients willing to sign written informed consent form
* Patients who meet the criteria for the first cross-sectional investigation and have an HbA1c < 7% will receive the second cross-sectional investigation

Exclusion Criteria:

* Patients unable or unwilling to comply with the requirements of the protocol

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 833 (Actual)
Dates: Start 2010-05-31 (Actual); Primary Completion 2012-03-31 (Actual); Study Completion 2012-03-31 (Actual)

PRIMARY OUTCOMES:
HbA1c change between the baseline and end of study | From baseline to month 6
Successful rate of blood glucose control (the proportion of patients with HbA1c <7%) | From baseline to month 6

SECONDARY OUTCOMES:
SMBG frequency change between the baseline and the end of the study | From baseline to month 6
Relationship between SMBG frequency change and blood glucose control | From baseline to month 6
To evaluate the change of quality of life in the 6 months by the health questionnaire SF-36 | From baseline to month 6

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Petersen, Study Director — Roche Diagnostics (Shanghai) Ltd
Locations (10):
- China (10):
  - Beijing
  - Chengdu
  - Guangzhou
  - Hangzhou
  - Nanjing
  - Shanghai
  - Shenyang
  - Tianjin
  - Wuhan
  - Xi'an